CLINICAL TRIAL: NCT04711421
Title: Using Pedometers for the Assessment and Enhancement of Mobility in Gynaecological and Oncological Patients Following Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 0689-19
Record Dates: First submitted 2021-01-09; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-05

CONDITIONS: Surgery; Mobilization; Gynecologic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Feedback (Experimental): Patients in this arm will wear a pedometer following gynecology and gynecology oncology surgeries until discharge. During this period, they will recieve feedback regrding the number of steps taken by them at the end of each day
  Interventions: Device: 4 VIVOFIT-
- No Intervention: Control (No Intervention): Patients in this arm will wear a pedometer following gynecology and gynecology oncology surgeries until discharge. During this period, they will recieve no feedback regrding the number of steps taken by them.

INTERVENTIONS:
Device: 4 VIVOFIT- — Feedback on number of steps taken by patint, as recorded by pedometers, provided by research team
  Arms: Experimental: Feedback

SUMMARY:
This is a prospective cohort study, planned to study the effects of pedometers (digital step counters) on patient mobility following gynecology and gynecology oncology surgeries. The investigators plan to study the effect of personalized repeated feedback approach based on pedometer results in patients following gynecology and gynecology oncology surgeries.

ELIGIBILITY:
Inclusion Criteria:

Patients following gynecology and gynecology oncology surgery Consent to participation No medical recommendation for bed rest and limited mobility

Exclusion Criteria:

Refusal to participate Medical recommendation to limit mobility

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of steps per day during the hospitalization period | Up to 1 week
  umber of steps taken by patient as recirded by pedometer

SECONDARY OUTCOMES:
Number of participants with complication following surgery | Up to 1 week
  infectious ( wound), blood product transfusion
Number of analgesic doses | Up to 1 week
  Number of doses of analgesics consumed by patient
Length of hospitalization | Up to 4 week
  Duration of hospitalization following surgery
Number of thromboembolic events | Up to 4 week
  hromboembolic events, including deep vein thrombosis and pulmonary emboli

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganer Herman H, Kleiner I, Tairy D, Gonen N, Ben Zvi M, Kovo M, Bar J, Weiner E. Effect of Digital Step Counter Feedback on Mobility After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2020 Jun;135(6):1345-1352. doi: 10.1097/AOG.0000000000003879. PMID 32459426